CLINICAL TRIAL: NCT05166746
Title: A Double-blind, Placebo-controlled Multicenter Trial on the Effect of Clindamycin and a Live Biotherapeutic on the Reproductive Outcomes of IVF Patients With Abnormal Vaginal Microbiota
Brief Title: The Effect of Clindamycin and a Live Biotherapeutic on the Reproductive Outcomes of IVF Patients With Abnormal Vaginal Microbiota
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, MD, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVM_Lacto_2015/582
Record Dates: First submitted 2021-08-24; First posted 2021-12-22 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Bacterial Vaginoses; Infertility, Female
MeSH Terms: conditions — Vaginosis, Bacterial; Infertility, Female | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Moreover, an interim analysis will be performed by blinded outcomes assessors according to the primary outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Clindamycin + LACTIN-V (L.crispatus) (Active Comparator): Oral Clindamycin 300 mg 2 times per day for 7 days followed by LACTIN-V (Osel, Inc.) until completion of the clinical pregnancy scan at week 7-9.
  Interventions: Drug: Clindamycin
- Clindamycin + placebo LACTIN-V (Active Comparator): Oral Clindamycin 300 mg 2 times per day for 7 days followed by LACTIN-V placebo (Osel, Inc.) until completion of the clinical pregnancy scan at week 7-9.
  Interventions: Drug: Clindamycin
- Placebo clindamycin + placebo LACTIN-V (Placebo Comparator): Matching clindamycin placebo 2 times per day for 7 days followed by LACTIN-V placebo (Osel Inc.) until completion of the clinical pregnancy scan at week 7-9.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clindamycin — Oral clindamycin 300mg/2xdaily in 7 days. LACTIN-V applicators 1x at night in 7 days, then 2xper week at night for 7 weeks.
  Other Names: LACTIN-V
  Arms: Clindamycin + LACTIN-V (L.crispatus); Clindamycin + placebo LACTIN-V
Other: Placebo — The Clindamycin placebo appear identical to active clindamycin by filling capsules with Mannitolium.
  The LACTIN-V placebo product has no intrinsic effect and is used to study the effect of the therapeutically active product. It is supplied as a pre-filled vaginal applicator packaged under nitrogen gas with one desiccant packet (0.25 g) in a sealed foil pouch. Each applicator contains 200 mg of LACTIN-V placebo powder containing the inactive ingredients of the LACTIN-V drug product, but not Lactobacillus crispatus CTV-05 (CTV-05), the active ingedient. The excipients used in the manufacture of LACTIN-V placebo are identical to those in the LACTIN-V drug product. Each placebo applicator contains the following constituents: maltodextrin, trehalose, xylitol, colloidal silicon dioxide, and sodium ascorbate
  Arms: Placebo clindamycin + placebo LACTIN-V

SUMMARY:
Study question: Does antibiotic alone or in combination with live biotherapeutic treatment of an abnormal vaginal microbiota improve the reproductive outcomes of IVF couples?

Study hypothesis:

The investigator hypothesize that treatment of the reproductive tract pathogens and restoration of vaginal Lactobacillus will improve the reproductive outcomes of IVF patients.

What is known already? Ultra-deep sequencing methods enable the refinement of reproductive tract microbiology in infertile patients. A recent meta-analysis reported that 19% of infertile patients had abnormal vaginal microbiota Moreover, someone have detected the presence of a Gardnerella (G.) vaginalis dominated endometrial biofilm in 50% of non-infertile patients with abnormal vaginal microbiota undergoing curettage; thus the treatment of such an endometrial biofilm might play an important role for the endometrial receptivity and subsequently the clinical pregnancy rate.

Pilot study: In a recent pilot study it was observed that an abnormal vaginal microbiota negatively affects the clinical pregnancy rate in IVF patients. In this study the prevalence of abnormal vaginal microbiota was 28% (36/130) and only 9% of patients with qPCR defined abnormal vaginal microbiota obtained a clinical pregnancy (p=0.004). This association remained significant in an adjusted analysis. Furthermore, the invetigators have preliminary results demonstrating that vaginal bacteria such as G. vaginalis can be found in the endometrium of IVF patients, which is also supported by recent publications

What is the novelty of this study? To the investigators knowledge, no previous treatment study of abnormal reproductive tract microbiota has been performed in IVF patients; this relatively small intervention holds the potential to increase the baby-take-home rate after IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal vaginal microbiota.
* The screening swab should be repeated if more than 3 months old.
* HIV, Hepatitis B or C positivity.
* First, second or third IVF stimulation cycle or embryo transfer therefrom.
* BMI<35
* Written informed consent.

Exclusion Criteria:

* Known or suspected hypersensitivity to clindamycin.
* HPV CIN 2 or higher.
* Former or current inflammatory bowel disease
* Severe concomitant disease, including diabetes.
* MAX 2 embryos may be transferred
* Artificial heart valve
* Intrauterine malformations with operation indication as determined by treating physician (Polyps, Septum, fibroma)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Estimated)
Dates: Start 2017-12-07 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy per embryo transfer | 7-9 weeks
  Ultrasound scan detection of intrauterine fetal heartbeat in gestational week 7-9

SECONDARY OUTCOMES:
Cure of abnormal vaginal microbiota | 1-2 months
  A vaginal swab and qPCR-validated diagnostics for abnormal vaginal microbiota
Live birth rate | 25-42 weeks depending on pregnancy.
  The birth of a live born child after 25 gestational weeks.
Biochemical pregnancy | 14 days gestation
  positive hCG blood test
Implantation rate | pregnancy scan at 7-9 weeks
  The number of embryos implanting
early miscarriage | 14 days - 12 weeks gestation
  The loss of an hCG positive pregnancy
Number of late miscarriage | 12 weeks gestation - to labour (i.e. not including still birth)
  The of pregnancy in late pregnancy
Number of preterm birth | prior to 37 gestational weeks
  birth of a liveborn
Birth weight | 25-42 weeks gestation depending on pregnancy
  weight at birth

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Stork Fertility Clinic VivaNeo, Copenhagen
  - Hvidovre Hospital, The Fertility Clinic, Hvidovre
  - Fertility Clinic Skive, Skive Regional Hospital, Skive

IPD SHARING:
Plan to Share IPD: Undecided
To this date, the Danish Data Protection agency does not allow IPD to be shared. But if possible we will do so.